CLINICAL TRIAL: NCT06669845
Title: Prospective Study of the Variation in the Angle of Anteflexion of the Uterus Before and After Micturition in Nulliparous Women With Uterine Anteversion.
Acronym: FLEXIMIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC24.0124; 2024-A01255-42 (Other: ANSM)
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-02

CONDITIONS: Uterine Anteflexion
Keywords: Uterine anteflexion; Nulliparous women; Full bladder; Ultrasound measurements
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ultrasonography pelvic (Other): Ultrasound measurements before and after bladder emptying
  Interventions: Procedure: Ultrasonography, Pelvic

INTERVENTIONS:
Procedure: Ultrasonography, Pelvic — Ultrasound measurements will be taken before and after bladder emptying. The axes of the uterine body, cervix and vagina will be marked out by tracing the 3 corresponding lines on the image.

SUMMARY:
A monocentric, prospective, comparative, and descriptive clinical study examining the uterine anteflexion angle before and after bladder emptying in nulliparous women with uterine anteversion. The study aims to assess how bladder fullness affects the anteflexion angle, which may impact the ease of intrauterine device (IUD) insertion. The primary objective is to determine the variation in the angle of anteflexion of the uterus before and after micturition in nulliparous women with uterine anteversion. Ultrasound measurements will be taken before and after bladder emptying. A secondary objective is to determine the prevalence of uterine anteversion in nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over;
* Nulliparous ;
* Feeling the need to urinate;
* Affiliated to a Social Security scheme.

Exclusion Criteria:

* Pregnant women;
* Desire of pregnancy with conception in progress;
* Primary amenorrhea ;
* Menopause ;
* Previous surgical termination of pregnancy;
* Previous medical abortion;
* Previous hysterectomy ;
* Previous conization;
* Absence of uterus;
* Irrepressible need to urinate;
* Inability or refusal to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
To determine the variation in the angle of anteflexion of the uterus before and after micturition in nulliparous women with uterine anteversion. | 1 day
  Difference between mean uterine anteflexion angle full bladder and empty bladder in nulliparous women with uterine anteversion.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement